CLINICAL TRIAL: NCT06890481
Title: Collaborative Development of a Virtual Reality Scenario, Integrated Into a Robotic Upper Limb Rehabilitation Device, for the Treatment of Unilateral Spatial Negligence (NSU) Through Mutisensory Stimulation: Feasibility and Usability Pilot Study
Brief Title: Robotic rEhabilitation sCenario fOr patieNts With NeglECT
Acronym: RECONNECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Humanware S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECONNECT
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Ischemic Stroke; Haemorrhagic Stroke; Neglect, Hemispatial
Keywords: stroke; robotics; end-effector; upper-limbs; rehabilitation; neglect; usability
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Perceptual Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Upper limbs robotic intervention (Experimental): The intervention, which includes the upper limb robotic device MOTORE+ and the new scenario, consists of:
  * Enrollment (Session 1): assessment of the inclusion criteria. Informed consent is obtained.
  * Baseline evaluation (Session 2): assessment of upper limb function and hemi-inattention. Additionally, robotic performance parameters are collected.
  * Training sessions (Sessions 3-12): these are the actual training sessions with the robotic device. Each session consists of three phases.
  In the first phase, the therapist provides the patient with the necessary information for the session.
  In the second phase, patients complete a pre-scenario session, during which the robotic parameters are adjusted.
  In the third phase, the scenario is used for motor and cognitive training.
  -Final evaluation (Session 13): final functional, clinical, and psychological assessments.
  The sessions are conducted five times per week, each lasting 45 minutes.
  Interventions: Device: Upper-limb planar robotic intervention

INTERVENTIONS:
Device: Upper-limb planar robotic intervention — The training sessions consist of three phases.
  In the first, the therapist provides the patient with the necessary information for the session.
  In the second, patients undergo a pre-scenario phase, in which the parameters of the robot (ratio between virtual and physical space, viscosity, and weight) are adjusted.
  In the third phase, the scenario is used for motor and cognitive exercise.
  Specifically, the scenario consists of a reaching exercise involving sequential stimuli placed in different spatial areas. The scenario has adaptive characteristics regarding:
  * Type of stimuli
  * Size of the stimuli
  * Visual and auditory cues
  * Number of stimuli, related to the space in which they are displayed.
  Each of these characteristics is adjusted differently according to the scenario's difficulty level. Regardless of the difficulty level, the scenario provides assistance as needed through a guided path (both visual and movement-based) toward the target.

SUMMARY:
The goal of this pilot clinical trial is to develop an integrated motor and cognitive rehabilitation program and evaluate the usability and acceptability of a new virtual reality scenario designed for the MOTORE device. This study will focus on the rehabilitation of the upper limbs in post-stroke patients with plegia and left-sided hemi-inattention. The main questions it aims to answer are:

* The evaluation of the usability and acceptability of the newly developed scenario
* The evaluation of the effects of the new scenario on patients' hemi-inattention
* The evaluation of changes in upper limb functional parameters

Participants will undergo a total of 13 rehabilitation sessions, each lasting 45 minutes, using the new scenario, including an initial and final assessment.

DETAILED DESCRIPTION:
Stroke in the right hemisphere can provoke both motor and cognitive symptoms. Hemi-inattention is a cognitive deficit typical of right hemispheric damage, with an incidence ranging from 12% to 95%. This deficit can manifest as difficulty in detecting and responding to stimuli from the left side of space, without any motor or sensory impairments that could justify the deficit. Hemi-inattention is usually associated with lesions in the inferior and superior parietal areas and, sometimes, in parts of the frontal area and the white matter connecting the parietal to the prefrontal areas. Hemi-inattention significantly compromises patients' quality of life and can negatively impact both motor and cognitive rehabilitation outcomes.

According to the theory of premotor spatial attention, brain attention and motor circuits are closely connected. Thus, it is possible to hypothesize that somatosensory activation in the contralesional space could stimulate the neural networks responsible for spatial representation and the conscious perception of stimuli. Some studies have attempted to verify this hypothesis by developing ad-hoc rehabilitation programs based on these theoretical principles. These studies can be divided into:

Studies investigating upper limb active mobilization, which require the activation of residual motor capabilities Studies investigating upper limb passive mobilization. It is widely accepted that hemi-inattention is a multisensory deficit, i.e., involving several sensory channels, and that a rehabilitation program based on joint stimulation of different channels can be effective.

Robot-assisted rehabilitation for the upper limbs, especially in hemiparetic patients, has gained growing interest in recent years, given the possibility of intensive treatment while still ensuring patient safety [8-9]. However, few studies have focused on the use of robotic devices, whose training modality often involves serious games, on cognitive aspects, particularly on hemi-inattention.

Even though preliminary and based on small sample sizes, these studies suggest a potential advantage of integrated cognitive and motor intervention for the rehabilitation of the upper limb and hemi-inattention. Indeed, the use of serious games and virtual reality scenarios can promote a synergistic effect of motor and cognitive stimulation. Furthermore, robotic rehabilitation can offer additional advantages, such as the "game effect," the ability to adapt the exercise difficulty level to the patient's performance, and the possibility of providing real-time feedback to the patient.

MOTORE is a planar end-effector robot for upper limb rehabilitation. In the literature, studies on the efficacy of this device in improving speed, strength, and spasticity of the upper limbs are available. However, no evidence is available regarding its use in treating hemi-inattention in post-stroke patients.

For this reason, this study aims to extend the use of the MOTORE device to the cognitive domain by creating a new virtual reality scenario for the robot. The scenario will consist of a sequential visual stimuli exercise with intra-session adaptive difficulty, designed to guide the patient's attention toward the neglected side of space through the combined use of visual and auditory stimuli and motor requests. The new scenario will be evaluated for usability with plegic post-stroke patients suffering from left hemi-inattention.

The novelty of the current study lies in the application of a multisensory approach, using auditory and visual stimuli, along with movement supported by the robot, to direct the patient's attention to the stimulus placed on the side of space affected by hemi-inattention.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a diagnosis of right hemispheric stroke
* Presence of a diagnosis of hemi-inattention (Apple test)
* Presence of left hemiplegia (Fugl-Meyer Assessment Upper Limb ≤58)
* Adjusted Montreal Cognitive Assessment <20
* Written informed consent

Exclusion Criteria:

* Presence of cognitive decline prior to the event
* Presence of previous stroke events
* Presence of osteoarticular rigidity (e.g., ankylosis, functional limitations with traumatic or degenerative origin) or spasticity in the affected upper limb (Modified Ashworth Scale ≥3 on shoulder, elbow, or wrist)
* Inability to maintain a sitting position
* Presence of severe visual disabilities
* Recent injection of botulinum toxin in the upper limb or planned injection of botulinum toxin during the study period
* Orthopaedic, neurological, or psychiatric disorders that could interfere with the study procedures and motor or cognitive assessments
* Unstable fractures of the upper limb
* Severe osteoporosis
* Skin lesions on the upper limb

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Usability of the device | Evaluated at session 12 (after the treatment) at an average of 2 weeks
  System Usability Scale (SUS)
Acceptability of the device for the operator | Evaluated at session 12 (after the treatment) at an average of 2 weeks
  Self-designed qualitative checklist

SECONDARY OUTCOMES:
Variation of symptoms connected to hemi-inattention | Evaluated at session 2 (before the beginning of treatment) and at session 12 (after treatment)
  Apple test
Functional direct effect of the device | Evaluated at session 2 (before the beginning of treatment) and at session 12 (after treatment)
  Fugl-Meyer Assessment for Upper Limbs

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi onlus, Florence, Firenze, Italy

REFERENCES:
- [Background] Robertson, I. H., & Hawkins, K. (1999). Limb activation and unilateral neglect. Neurocase, 5(2), 153-160
- [Background] Heilman, K. M., Watson, R. T., & Valenstein, E. (1993). Neglect and related disorders. In K. M. Heilman & E. Valenstein (Eds.), Clinical neuropsychology (pp. 279-336). Oxford University Press.
- [Background] Rizzolatti G, Berti A. Neglect as a neural representation deficit. Rev Neurol (Paris). 1990;146(10):626-34. PMID 2124720
- [Background] Robertson, I. H., Hogg, K., & McMillan, T. M. (1998). Rehabilitation of unilateral neglect: improving function by contralesional limb activation. Neuropsychological rehabilitation, 8(1), 19-29
- [Background] Gainotti G, Perri R, Cappa A. Left hand movements and right hemisphere activation in unilateral spatial neglect: a test of the interhemispheric imbalance hypothesis. Neuropsychologia. 2002;40(8):1350-5. doi: 10.1016/s0028-3932(01)00211-1. PMID 11931938
- [Background] Frassinetti F, Rossi M, Ladavas E. Passive limb movements improve visual neglect. Neuropsychologia. 2001;39(7):725-33. doi: 10.1016/s0028-3932(00)00156-1. PMID 11311302
- [Background] Jacobs S, Brozzoli C, Farne A. Neglect: a multisensory deficit? Neuropsychologia. 2012 May;50(6):1029-44. doi: 10.1016/j.neuropsychologia.2012.03.018. Epub 2012 Mar 28. PMID 22465475
- [Background] Mehrholz J, Pollock A, Pohl M, Kugler J, Elsner B. Systematic review with network meta-analysis of randomized controlled trials of robotic-assisted arm training for improving activities of daily living and upper limb function after stroke. J Neuroeng Rehabil. 2020 Jun 30;17(1):83. doi: 10.1186/s12984-020-00715-0. PMID 32605587
- [Background] Bertani R, Melegari C, De Cola MC, Bramanti A, Bramanti P, Calabro RS. Effects of robot-assisted upper limb rehabilitation in stroke patients: a systematic review with meta-analysis. Neurol Sci. 2017 Sep;38(9):1561-1569. doi: 10.1007/s10072-017-2995-5. Epub 2017 May 24. PMID 28540536
- [Background] Varalta V, Picelli A, Fonte C, Montemezzi G, La Marchina E, Smania N. Effects of contralesional robot-assisted hand training in patients with unilateral spatial neglect following stroke: a case series study. J Neuroeng Rehabil. 2014 Dec 5;11:160. doi: 10.1186/1743-0003-11-160. PMID 25476507
- [Background] Choi YS, Lee KW, Lee JH, Kim SB, Park GT, Lee SJ. The Effect of an Upper Limb Rehabilitation Robot on Hemispatial Neglect in Stroke Patients. Ann Rehabil Med. 2016 Aug;40(4):611-9. doi: 10.5535/arm.2016.40.4.611. Epub 2016 Aug 24. PMID 27606267
- [Background] Heins, S., Dehem, S., Montedoro, V., Dehez, B., Edwards, M., Stoquart, G., ... & Lejeune, T. (2017, April). Robotic-assisted serious game for motor and cognitive post-stroke rehabilitation. In 2017 IEEE 5th International Conference on Serious Games and Applications for Health (SeGAH) (pp. 1-8). IEEE.
- [Background] Mazzoleni S, Battini E, Crecchi R, Dario P, Posteraro F. Upper limb robot-assisted therapy in subacute and chronic stroke patients using an innovative end-effector haptic device: A pilot study. NeuroRehabilitation. 2018;42(1):43-52. doi: 10.3233/NRE-172166. PMID 29400670